CLINICAL TRIAL: NCT06678594
Title: Implementation of a Standardized Algorithm for CoronarY CaLcificatiOn With PlaquE Modification Using UltraSound Guidance to Improve Procedural and Clinical Outcomes (CYCLOPES)
Brief Title: Implementation of a Standardized Algorithm for Coronary Calcification With Plaque Modification
Acronym: CYCLOPES
Status: Recruiting | Type: Observational
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Cardiovascular Research Institute Dublin (Other)
Responsible Party: Sponsor
Other Study IDs: CYCLOPES V1.1
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Myocardial Ischaemia; Severely Calcified Coronary Stenoses; Coronary Calcification
Keywords: calcium modification; coronary calcification; plaque modification; IVUS; Intravascular Ultrasound; calcium modification algorithm
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient treatment will follow a standardised algorithm for calcium modification: All patients will have coronary angiography (QCA) and intravascular ultrasound (IVUS) imaging with 60MHz HD IVUS of the calcified lesion at baseline. The lesion will be characterized based on calcium distribution and morphology as assessed by HD IVUS. Depending on the specific lesion characteristics, the appropriate method for calcium modification will be chosen and performed in line with the CYCLOPES calcium modification algorithm included in the study protocol.
  The calcific lesion will be imaged for a second time by 60MHz HD IVUS following calcium modification. The operator will then proceed, if no further lesion preparation is required, to deploy a bioabsorbable polymer Everolimus eluting stent using standard stenting techniques, post dilatation will be performed at the operator's discretion. The treated lesion will be assessed again using intravascular ultrasound following stent deployment and optimization.
  Interventions: Procedure: Calcium modification

INTERVENTIONS:
Procedure: Calcium modification — Patients will undergo one or more of the following procedures, subject to the algorithm:
  Angioplasty Balloon Cutting Balloon Rotational Atherectomy Intravascular Lithotripsy
  Other Names: plaque modification

SUMMARY:
In this study, the doctors will follow a set of rules that is called an algorithm. An algorithm is a step-by-step approach that doctors use to guide them when making decisions about the best way to treat their patients. Algorithms are useful because they help doctors decide on the best treatment approach based on the patient's individual circumstances and the best medical evidence available. The algorithm that is being used in this study is called a calcium modification algorithm and it will guide doctors when deciding on the best way to modify or break up the calcium in coronary arteries.

In this study, we aim to prove that the calcium modification algorithm, described above, safely and effectively guides doctors on the best way to modify calcium in patients' coronary arteries. By doing so, it will help doctors in making decisions about patients' treatment during their procedure. It will also help standardise care for patients, so patients receive the same treatment no matter what hospital they are in or what doctor is treating them.

DETAILED DESCRIPTION:
Investigational strategy:

Calcium modification algorithm to guide coronary intervention with an High Definition Intra Vascular Ultrasound (HD IVUS) imaging guided pathway that provides a systematic approach to coronary modification.

Objectives:

The aim of this study is to validate a comprehensive and intravascular imaging-based calcium modification algorithm for the treatment of moderate to severely calcified coronary lesions.

Study Population:

Patients with coronary artery disease with evidence of moderate to severely calcified coronary arterial lesions that are planned for percutaneous intervention requiring calcium modification.

Design:

CYCLOPES is a prospective, multicenter, open-label, single arm trial assessing the feasibility and efficacy of an intracoronary ultrasound guided algorithm for calcium modification in patients undergoing percutaneous coronary intervention (PCI) for chronic calcific coronary artery disease. The study will enrol 500 patients who will undergo PCI with calcium modification.

Participants will be enrolled prospectively in 25 sites in Ireland, Switzerland, the United Kingdom, Spain, France, Italy and Germany (7 countries).

All patients will have coronary angiography (QCA) and intravascular ultrasound (IVUS) imaging with 60MHz HD IVUS of the calcified lesion at baseline. The lesion will be characterized based on calcium distribution and morphology as assessed by HD IVUS. Depending on the specific lesion characteristics, the appropriate method for calcium modification will be chosen and performed in line with the CYCLOPES calcium modification algorithm included in the study protocol.

The calcific lesion will be imaged for a second time by 60MHz HD IVUS following calcium modification. The operator will then proceed, if no further lesion preparation is required, to deploy a bioabsorbable polymer Everolimus eluting stent using standard stenting techniques, post dilatation will be performed at the operator's discretion. The treated lesion will be assessed again using intravascular ultrasound following stent deployment and optimization.

The primary end points will be the post stenting minimal stent area (MSA) at the site of maximum calcification relative to reference lumen area assessed with 60MHz HD IVUS and target lesion failure (TLF) at 1-year post-procedure. All HD IVUS determined endpoints will be assessed at an independent imaging core laboratory.

Participants will be assessed with clinic or phone visits at hospital discharge, 1 month and 12-month time points post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Documented myocardial ischaemia.
2. At least one moderate to severely calcified native coronary artery lesion confirmed by QCA and/or 60MHz HD IVUS, with the presence of significant calcium, ≥70% diameter stenosis by visual estimation (in a reference vessel diameter of ≥2.5mm and ≤4.0mm) and TIMI 3 flow at baseline that is suitable for PCI.

   a. Significant calcium at the target lesion site is defined as either: i. The presence of radiopacities involving both sides of the arterial wall >10mm and involving the target lesion on angiography.

   or ii. The presence of >270° arc of superficial calcium on HD intravascular imaging with a length >5mm or the presence of 360° arc of calcium on HD intravascular imaging. [1]
3. It is possible to cross the calcified lesion with a coronary guidewire.
4. Age ≥ 18 years.
5. Patient is willing and able to comply with the study procedures and follow-up.

Exclusion Criteria:

1. Patients with cardiogenic shock.
2. ST-segment elevation myocardial infarction.
3. Instent re-stenosis.
4. Stent thrombosis.
5. Coronary artery dissection.
6. Chronic total occlusion in a major artery.
7. Left ventricular ejection fraction ≤30%. Need for coronary artery bypass graft surgery.

9. Documented allergy to everolimus or to any stent material 10. Any contraindication for dual antiplatelet therapy with aspirin and a P2Y12 inhibitor for at least 3 months (except for patients on oral anticoagulation). 11. For female, pregnancy, breastfeeding or intend to become pregnant within 1 year 12. Life expectancy <1 year. 13. Participation in another study with an investigational product. 14. Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe coronary calcification requiring calcium modification and percutaneous coronary revascularization
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2026-03-23 (Estimated); Study Completion 2027-03-23 (Estimated)

PRIMARY OUTCOMES:
Minimum stent area (MSA) | End of Index Procedure
  Minimum stent area (MSA) at the site of maximum calcification measured at the end of the index procedure
Target lesion failure (TLF) | At Year 1
  Target lesion failure (TLF) (cardiovascular death, non-fatal myocardial infarction (MI) related to the target vessel, unplanned ischemia-driven target lesion revascularization) at 1 year

SECONDARY OUTCOMES:
Individual components of TLF at 1 month and 1 year | At 1 month and 1 year
  Individual components of TLF at 1 month and 1 year
Minimum stent area (MSA) at the end of the index procedure | At end of index procedure
  Minimum stent area (MSA) at the end of the index procedure
Strategy Success | At end of index procedure
  Strategy success defined as:
  1. Successful stent delivery
  2. ≥ 80% stent expansion
  3. Complete stent apposition
  4. No edge dissection
  5. Full lesion coverage with <50% plaque burden at proximal and distal references
  6. TIMI 3 flow
Target vessel revascularization (TVR) | At Year 1
  Target vessel revascularization (TVR)
Target lesion revascularization (TLR) | At Year 1
  Target lesion revascularization (TLR)
Stent thrombosis | At Year 1
  Stent thrombosis
Stroke | At Year 1
  Stroke
Cardiovascular death | At Year 1
  Cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Byrne, Principal Investigator — RCSI University of Medicine and Health Sciences
Locations (1):
- Mater Private Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, the study team plan to make anonymized study data available to members of the research community, both academic and industry, who request access to it. This is called open access to clinical trial data and the aim is to help other researchers and encourage transparency in clinical research by allowing other researchers 'test' the findings from this study and develop tools to help treatment of other patients in the future. Personal data will not be shared with anyone outside of those listed in the Patient Information Leaflet (ie Hospital Study Team, Members of committee monitoring the safety of the trial, sponsor auditor & regulatory authorities etc. It will not be possible to identify an individual as the data shared will be anonymized data, for example in addition to personal data being replaced by coding, date of birth with be changed to a date range (e.g. 35-44 yrs old) to ensure that patients cannot be identified from the data shared.

REFERENCES:
- [Derived] O'Callaghan D, Durand R, Hanratty CG, Cuisset T, Vaquerizo B, Sinning JM, O'Kane P, Coughlan JJ, Walsh S, Colleran R, Rai H, Soliman O, Barbato E, Stahli BE, Byrne RA. A Prospective, Multicenter, Open Label Study Investigating the Implementation of a Standardized Algorithm for Coronary CaLcificatiOn With PlaquE Modification Using UltraSound Guidance to Improve Procedural and Clinical Outcomes (CYCLOPES): Design and Rationale of the CYCLOPES Trial. Catheter Cardiovasc Interv. 2025 Dec 17. doi: 10.1002/ccd.70424. Online ahead of print. PMID 41408534

DOCUMENTS (1):
  • Study Protocol (2024-08-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT06678594/Prot_000.pdf